CLINICAL TRIAL: NCT01358734
Title: A Phase 2, Multicenter, Randomized, Open-label, Parallel-group Study of a Lenalidomide (Revlimid®) Regimen or a Sequential Azacitidine (Vidaza®) Plus Lenalidomide (Revlimid®) Regimen Versus an Azacitidine (Vidaza®) Regimen for Therapy of Older Subjects With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: A Study Being Conducted at Multiple Locations to Compare Safety and Efficacy of Three Different Regimens; (1) High-Dose Lenalidomide; (2) Lenalidomide + Azacitidine; or (3) Azacitidine in Subjects ≥ 65 Years With Newly-Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-AML-001
Record Dates: First submitted 2011-05-19; First posted 2011-05-24 (Estimated); Results first posted 2016-07-04 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Acute Myeloid Leukemia; Acute Myelogenous Leukemia
Keywords: AML; elderly; acute myelogenous leukemia; vidaza; azacitidine; elderly AML; revlimid; lenalidomide
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lenalidomide in combination with azacitidine (Experimental): Repeated cycles of azacitidine 75 mg/m^2/day subcutaneous (SC) on Days 1-7 and lenalidomide 50 mg/day by mouth (PO) on Days 8-28 followed by a 14-day break plus best supportive care
  Interventions: Drug: Azacitidine; Drug: Lenalidomide; Other: Best Supportive Care (BSC)
- Lenalidomide - single agent (Experimental): Lenalidomide 50 mg PO daily for 28 days for the first 2 cycles and lenalidomide 25 mg daily for 28 days for the next 2 cycles followed by continuous 28-day cycles of lenalidomide 10 mg daily PO plus best supportive care
  Interventions: Drug: Lenalidomide; Other: Best Supportive Care (BSC)
- Azacitidine-single agent (Experimental): Repeated cycles of azacitidine 75mg/m^2/day subcutaneous on Days 1-7 followed by a 21-day break plus best supportive care
  Interventions: Drug: Azacitidine; Other: Best Supportive Care (BSC)

INTERVENTIONS:
Drug: Azacitidine — Azacitidine at 75 mg/m^2/day subcutaneous on Days 1-7
  Other Names: Vidaza
  Arms: Azacitidine-single agent; Lenalidomide in combination with azacitidine
Drug: Lenalidomide — Lenalidomide 50 mg PO daily x 28 days for the first 2 cycles then 25 mg PO daily x 28 days for the next 2 cycles followed by continuous 28-day cycles of lenalidomide 10 mg PO daily
  Other Names: Revlimid®; CC-5013
  Arms: Lenalidomide - single agent; Lenalidomide in combination with azacitidine
Other: Best Supportive Care (BSC) — The use of BSC was considered as concomitant treatment and must be documented as concomitant medication.
  BSC includes, but is not limited to, treatment with Red Blood Celll (RBC) or whole blood transfusions, fresh frozen plasma transfusions, platelet transfusions, antibiotic or antifungal therapy, and nutritional support

SUMMARY:
The study aim is to compare safety and efficacy of high-dose lenalidomide regimen, sequential azacitidine and lenalidomide and an azacitidine in persons ≥65 years with newly-diagnosed acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
On September 11, 2013, randomization into the continuous 50 mg lenalidomide only arm was temporarily suspended based on review of the data from the first 13 participants and a high rate of discontinuation (11/13 participants). The Data Monitoring Committee assessed the study data on September 20, 2013 and reported no safety concerns. The high rate of early discontinuation is inconsistent with the treatment duration required for testing the study primary endpoint of survival at one year. Consequently, Celgene has decided not to reopen the lenalidomide only arm.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed acute myeloid leukemia (AML), AML with antecedent hematologic disorder or therapy-related AML
* Male or female subjects aged ≥ 65
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* White blood cell (WBC) count ≤ 10 x 10⁹/L at screening

Exclusion Criteria:

* Previous treatment with azacitidine, decitabine, cytarabine or lenalidomide
* Previous cytotoxic or biologic treatment of any kind for AML or prior use of targeted therapy agents.
* Suspected or proven acute promyelocytic leukemia
* Prior bone marrow or stem cell transplantation
* Candidate for allogeneic bone marrow or stem cell transplantation
* AML antecedent hematologic disorder such as chronic myelogenous leukemia or myeloproliferative neoplasms
* Presence of malignant disease within the previous 12 months with exceptions

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-04-27 (Actual); Primary Completion 2015-05-19 (Actual); Study Completion 2018-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gale, MD, Study Director — Celgene
Locations (30):
- United States (24):
  - (210) University of Arizona Cancer Center, Tucson, Arizona
  - (180) University of California, San Diego, La Jolla, California
  - (240) Cedars-Sinai Medical Center, Los Angeles, California
  - (215) Hematology Oncology Medical Group, Orange, California
  - (130) UC Davis Medical Center, Sacramento, California
  - (200) Coastal Integrative Cancer Care, San Luis Obispo, California
  - (125) University of Stanford, Stanford, California
  - (115) University of Colorado Anschultz Cancer Center, Aurora, Colorado
  - (145) Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - (140) Rush University Medical Center, Chicago, Illinois
  - (185) The University of Kansas Cancer Center, Westwood, Kansas
  - (175) University Lousiville, Louisville, Kentucky
  - (195) Tulane University Hospital Tulane Cancer Center, New Orleans, Louisiana
  - (235) University of Minnesota, Minneapolis, Minnesota
  - (100) Washington University School of Medicine, St Louis, Missouri
  - (150) Billings Clinic, Billings, Montana
  - (165) Mount Sinai Medical Center New York, New York, New York
  - (160) The Western Pennsylvania Hospital- Cancer Institute, Pittsburgh, Pennsylvania
  - (205) Greenville Hospital System, Greenville, South Carolina
  - (120) Avera Cancer Institute, Sioux Falls, South Dakota
  - (230) Tennessee Oncology, PLLC, Nashville, Tennessee
  - (105) University of Texas Southwestern Medical Center Simmons Comprehensive Cancer Center, Dallas, Texas
  - (155) Cancer Care Centers of South Texas, San Antonio, Texas
  - (135) University of Wisconsin, Madison, Wisconsin
- Canada (6):
  - (402) Tom Baker Cancer Centre, Calgary, Alberta
  - (405) University of Alberta Hospital, Edmonton, Alberta
  - (401) Cancer Care Manitoba, Winnipeg, Manitoba
  - (403) Queen Elizabeth II Health Sciences Centre - VG Site, Halifax, Nova Scotia
  - (404) The Ottawa Hospital, Ottawa, Ontario
  - (400) Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Medeiros BC, McCaul K, Kambhampati S, Pollyea DA, Kumar R, Silverman LR, Kew A, Saini L, Beach CL, Vij R, Wang X, Zhong J, Gale RP. Randomized study of continuous high-dose lenalidomide, sequential azacitidine and lenalidomide, or azacitidine in persons 65 years and over with newly-diagnosed acute myeloid leukemia. Haematologica. 2018 Jan;103(1):101-106. doi: 10.3324/haematol.2017.172353. Epub 2017 Nov 2. PMID 29097499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at 25 sites in North America (Canada and the United States).
Pre-assignment Details: Participants were centrally randomized 1:1:1 and stratified by the Eastern Cooperative Oncology Group (ECOG) performance score (0 to 1 versus 2) and peripheral blood blast count (<1 versus ≥ 1 x 10^9/L).
Groups:
- Lenalidomide: Participants received lenalidomide 50 mg daily (QD) by mouth (PO) for 28 days for the first 2 cycles followed by 25 mg QD PO for 28 days for the next 2 cycles followed by continuous 28-day cycles of oral lenalidomide 10 mg daily plus BSC, including antibiotics and transfusions, at the investigator's discretion.
- Azacitidine Plus Lenalidomide: Participants received azacitidine 75 mg/m^2/ QD administered subcutaneously (SC) on Days 1 through 7 and lenalidomide 50 mg QD PO on days 8 through 28 followed by a 14-day rest period plus BSC
- Azacitidine: Participants received azacitidine 75mg/m^2 administered SC on days 1 through 7 followed by a 21-day rest period plus BSC
Period: Overall Study
Arm/Group | Lenalidomide | Azacitidine Plus Lenalidomide | Azacitidine
Started | 15 | 39 | 34
Safety Population | 14 (The safety population includes all participants who received at least one dose of study drug.) | 38 (The safety population includes all participants who received at least one dose of study drug.) | 32 (The safety population includes all participants who received at least one dose of study drug.)
Completed | 0 | 0 | 0
Not Completed | 15 | 39 | 34
Not completed — Adverse Event | 4 | 7 | 3
Not completed — Lack of Efficacy | 0 | 1 | 3
Not completed — Withdrawal by Subject | 1 | 6 | 3
Not completed — Death | 3 | 7 | 2
Not completed — Progressive Disease | 5 | 13 | 16
Not completed — Non-compliance with study drug | 0 | 0 | 1
Not completed — Other | 2 | 5 | 4
Not completed — Protocol Violation | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent To Treat (ITT) includes all randomized participants
Groups:
- Azacitidine + Lenalidomide: Participants received azacitidine 75 mg/m^2/ daily SC on Days 1 through 7 and lenalidomide 50 mg daily PO on Days 8 through 28 followed by a 14-day rest period plus best supportive care
- Total: Total of all reporting groups
Arm/Group | Lenalidomide | Azacitidine + Lenalidomide | Azacitidine | Total
Number analyzed (Participants) | 15 | 39 | 34 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.6 (5.47) | 75.5 (5.88) | 74.8 (4.96) | 75.97 (5.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 17 | 15 | 35
  Male | 12 | 22 | 19 | 53
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — The ECOG Scale of Performance Status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. It has scores ranging from 0 to 5 and these correlate with scores from Karnofsky Scales 0-100. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  Participants
    0 = (Fully Active) | 4 | 4 | 10 | 18
    1 = (Restrictive but ambulatory) | 9 | 28 | 17 | 54
    (Ambulatory but unable to work) | 2 | 7 | 6 | 15
    3 = (Limited self care) | 0 | 0 | 0 | 0
    4 = (Completely Disabled) | 0 | 0 | 0 | 0
    Missing | 0 | 0 | 1 | 1
Peripheral Blast Blood Count [Count of Participants; unit: Participants]
  <1 X 10^9L | 11 | 31 | 27 | 69
  ≥1 X 10^9L | 4 | 8 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Kaplan Meier Estimates for One Year Survival
Description: One-year survival rate was defined as all deaths within one year from the date of randomization. All others censored at the at year 1 or date of discontinuation
Time Frame: Up to 24 months
Population: ITT included all randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide | Azacitidine Plus Lenalidomide | Azacitidine
Number analyzed (Participants) | 15 | 39 | 34
months | 3.00 [1.18 to 11.93] | 9.61 [3.18 to 19.31] | 13.67 [6.75 to NA] — The Upper limit of the 95% Confidence Interval could not be estimated due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Lenalidomide vs Azacitidine Plus Lenalidomide; Test type: Superiority or Other; p = 0.119, Log Rank; Hazard Ratio (HR) = 1.789, 95% CI 2-sided [0.861 to 3.718]
Statistical Analysis 2: Comparison: Lenalidomide vs Azacitidine; Test type: Superiority or Other; p = 0.014, Log Rank; Hazard Ratio (HR) = 2.659, 95% CI 2-sided [1.214 to 5.822]
Statistical Analysis 3: Comparison: Azacitidine Plus Lenalidomide vs Azacitidine; Test type: Superiority or Other; p = 0.356, Log Rank; Hazard Ratio (HR) = 1.367, 95% CI 2-sided [0.704 to 2.653]

2. Secondary Outcome: Percentage of Participants With a Complete Response or Morphologic Incomplete Response.
Description: Based on IWG response criteria for AML. Complete remission (CR), morphologic complete remission (CR) was defined as < 5% bone marrow blasts, an absolute neutrophil count ≥ 1 x 10^9/L, platelets ≥100 x 10^9/L, and transfusion independence (no transfusions for 1 week prior to each assessment). No duration of these findings is required for confirmation of this response.
  Morphologic CR with incomplete blood count recovery (CRi) was defined as a morphologic complete remission but the ANC count may be <1 x 10^9/L and/or the platelet count may be <100 x 10^9/L. Because of a high rate of discontinuation in one of the investigational cohorts, secondary endpoints were not analyzed.
Time Frame: Complete Response or Morphologic Incomplete Response data not analyzed.
Population: Because of a high rate of discontinuation in one of the investigational cohorts, secondary endpoints were not analyzed.
Arm/Group | Lenalidomide | Azacitidine Plus Lenalidomide | Azacitidine
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Duration of Remission (DoR)
Description: Duration of remission was defined as the time from the date of CR or CRi until relapse. Because of a high rate of discontinuation in one of the investigational cohorts, secondary endpoints were not analyzed.
Time Frame: Duration of Remission (DoR) time frame not analyzed.
Population: Because of a high rate of discontinuation in one of the investigational cohorts, secondary endpoints were not analyzed.
Arm/Group | Lenalidomide | Azacitidine Plus Lenalidomide | Azacitidine
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Cytogenetic Complete Remission Rate (CRc)
Description: The CRc response category is comprised of the subset of participants who had abnormal cytogenetics at baseline and subsequently achieved CR during treatment in conjunction with a reversion to a normal karyotype. For the primary definition of CRc, a normal karyotype is defined as no clonal abnormalities after review of at least 10 metaphases using conventional cytogenetic techniques. Cytogenetic complete remission rate (CRc) 1) CR criteria met AND 2) Abnormal karyotype present at baseline AND 3) Reversion to normal karyotype at time of CR (based on ≥ 10 metaphases), where date of cytogenetic sample = date of BM sample used for the CR assessment. Because of a high rate of discontinuation in one of the investigational cohorts, secondary endpoints were not analyzed.
Time Frame: Cytogenetic Complete Remission timeframe was not analyzed.
Population: Because of a high rate of discontinuation in one of the investigational cohorts, secondary endpoints were not analyzed.
Arm/Group | Lenalidomide | Azacitidine Plus Lenalidomide | Azacitidine
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants With an Overall Response Rate (CR +CRi+ PR)
Description: Morphologic complete remission (CR) is defined as a leukemia-free state defined as less than 5% blasts in a one marrow aspirate with spicules and with at least 200 nucleated cells (there should be no blasts with auer rods) and ANC of ≥ 1 x 10^9/L, a platelet count ≥ 100 x 10^9/L, no transfusions for 1 week prior to each assessment. No duration of these findings is required for confirmation of this response. Morphologic complete remission with incomplete blood count recovery was defined as a morphologic complete remission but the ANC may be < 1 x 10^9/L and/or the platelet count may be < 100 x 10^9/L. Partial remission was defined as an ANC > 1 x 10^9/L and platelet count ≥ 100 x 10^9/L with a > 50% decrease in the percentage of bone marrow blasts to 5% to 25% (a blast count value of ≤ 5% may also be considered a partial remission if auer rods are present). Because of a high rate of discontinuation in one of the investigational cohorts, secondary endpoints were not analyzed.
Time Frame: Overall response rate time frame was not analyzed.
Population: Because of a high rate of discontinuation in one of the investigational cohorts, secondary endpoints were not analyzed.
Arm/Group | Lenalidomide | Azacitidine Plus Lenalidomide | Azacitidine
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization to the first observation of documented disease progression or death from any cause whichever occurred first. Because of a high rate of discontinuation in one of the investigational cohorts, secondary endpoints were not analyzed.
Time Frame: Progression-Free survival data and time frame was not analyzed.
Population: Because of a high rate of discontinuation in one of the investigational cohorts, secondary endpoints were not analyzed.
Arm/Group | Lenalidomide | Azacitidine Plus Lenalidomide | Azacitidine
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Event-Free Survival (EFS)
Description: EFS was defined as the interval from the date of randomization to the date of treatment failure, progressive disease, relapse after CR or CRi, or death from any cause, whichever occurred first. Because of a high rate of discontinuation in one of the investigational cohorts, secondary endpoints were not analyzed.
Time Frame: Event-Free survival time was not analyzed.
Population: Because of a high rate of discontinuation in one of the investigational cohorts, secondary endpoints were not analyzed.
Arm/Group | Lenalidomide | Azacitidine Plus Lenalidomide | Azacitidine
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Relapse-Free Survival (RFS)
Description: RFS is defined only for subjects that achieve CR and CRi and is measured as the interval from that date to the date of disease relapse, death from any cause, whichever occurs first, censoring at the last visit date for subjects alive in continuous CR/CRi. Because of a high rate of discontinuation in one of the investigational cohorts, secondary endpoints were not analyzed.
Time Frame: Relapse-Free survival time frame was not analyzed.
Population: Because of a high rate of discontinuation in one of the investigational cohorts, secondary endpoints were not analyzed.
Arm/Group | Lenalidomide | Azacitidine Plus Lenalidomide | Azacitidine
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Percentage of Participants With 30-Day Treatment-Related Mortality
Description: 30-day mortality rate was defined as death from any cause within 30 days after first dose.
Time Frame: 30 days
Population: ITT included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide | Azacitidine Plus Lenalidomide | Azacitidine
Number analyzed (Participants) | 15 | 39 | 34
percentage of participants | 13.3 | 17.9 | 5.9

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE)
Description: TEAEs were defined as those events that started on or after the first day of study drug up until 28 days after the last dose of study drug; Serious AE (SAE) = any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability; is a congenital anomaly/birth defect; constitutes an important medical event. Severity of AEs were graded based upon the participants symptoms according to the Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0); and according to the scale: Grade (Gr) 1 = Mild - transient or mild discomfort; no medical intervention required; Grade 2 = Moderate - mild to moderate limitation in activity; Grade 3 = Severe; Grade 4 = Life threatening; Grade 5 = Death
Time Frame: From the first dose of study drug up to 28 days after the last dose of study drug; up to 15 May 2018
Population: Safety population includes all participants who have received at least 1 dose of Investigational Product.
Measure: Number; unit: participants
Arm/Group | Lenalidomide | Azacitidine Plus Lenalidomide | Azacitidine
Number analyzed (Participants) | 14 | 38 | 32
participants
  Any TEAE | 14 | 38 | 32
  ≥1 TEAE related to study drug | 13 | 35 | 30
  ≥1 TEAE CTCAE Grade 3 or 4 TEAE | 14 | 34 | 29
  ≥1 TEAE CTCAE Gr 3 or 4 TEAE related to study drug | 11 | 25 | 18
  ≥1 TEAE CTCAE Grade 5 | 5 | 10 | 5
  ≥1 Serious TEAE | 13 | 29 | 25
  ≥1 Serious TEAE related to study drug | 10 | 16 | 7
  ≥1TEAE leading to discontinuation of study drug | 6 | 12 | 4
  ≥1TEAE leading to dose reduction of study drug | 0 | 8 | 2
  ≥1TEAE leading to dose interruption of study drug | 8 | 21 | 10

11. Other Pre Specified Outcome: Percentage of Participants Alive at One Year
Description: Defined as the percentage of participants who survived at one year
Time Frame: Up to 12 months
Population: ITT population included participants who were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenalidomide | Azacitidine Plus Lenalidomide | Azacitidine
Number analyzed (Participants) | 15 | 39 | 34
Percentage of participants | 21.4 [0.0 to 42.9] | 43.9 [27.9 to 59.9] | 52.3 [34.7 to 69.8]

12. Primary Outcome: Overall Survival
Description: Overall Survival reported at the end of the study are for those participants who were alive at the end of the study
Time Frame: From date of randomization until the date of the first documented date of progression or date of death of any cause; the overall median follow-up for survivng participants was 4.1 months (range 0.2 to 54.8 months)
Population: Participants who were still alive at the end of the study and in safety population.
Measure: Median (Full Range); unit: months
Arm/Group | Lenalidomide | Azacitidine Plus Lenalidomide | Azacitidine
Number analyzed (Participants) | 1 | 4 | 3
months | 0.2 [0.2 to 0.2] | 7.1 [1.4 to 53.3] | 4.1 [0.2 to 54.8]

13. Secondary Outcome: Number of Participants With a Second Primary Malignancy
Description: Second primary malignancies were monitored as events of interest and reported as serious adverse events regardless of the treatment arm the participant was enrolled in.
Time Frame: From randomization of the last participant up to a minimum of 4 years following discontinuation
Population: Safety population includes all participants who received at least one dose of IP
Measure: Number; unit: Participants
Arm/Group | Lenalidomide | Azacitidine Plus Lenalidomide | Azacitidine
Number analyzed (Participants) | 14 | 38 | 32
Participants | 0 | 0 | 3

ADVERSE EVENTS:
Time Frame: From the date of randomization to 28 days after the last dose of study drug. Up to 15 May 2018.
Description: Between the date of first dose of IP up until and 28 days after the date of last dose of IP or that were present prior to the first day of IP but increased in severity or were assessed as related to IP during the study, including the follow-up 28-day time interval. All-cause mortality includes all deaths that occurred during the entire study.
Arm/Group | Lenalidomide | Azacitidine Plus Lenalidomide | Azacitidine
All-Cause Mortality (participants affected / at risk) | 7/14 | 34/38 | 29/32
Serious Adverse Events (participants affected / at risk) | 13/14 | 29/38 | 25/32
Other Adverse Events (participants affected / at risk) | 14/14 | 38/38 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=14) | Azacitidine Plus Lenalidomide (N=38) | Azacitidine (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 16 | 8
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 4 | 7
Sepsis (Infections and infestations) | 2 | 1 | 2
Cellulitis (Infections and infestations) | 0 | 3 | 1
Septic shock (Infections and infestations) | 2 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 2
Klebsiella bacteraemia (Infections and infestations) | 0 | 2 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 1
Breast abscess (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1
Enterobacter bacteraemia (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 2 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Performance status decreased (General disorders) | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 2
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blast cell count increased (Investigations) | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Bone marrow myelogram abnormal (Investigations) | 0 | 0 | 1
Megakaryocytes decreased (Investigations) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 2 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Leukaemic infiltration extramedullary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=14) | Azacitidine Plus Lenalidomide (N=38) | Azacitidine (N=32)
Constipation (Gastrointestinal disorders) | 7 | 24 | 17
Nausea (Gastrointestinal disorders) | 4 | 19 | 22
Diarrhoea (Gastrointestinal disorders) | 5 | 19 | 8
Vomiting (Gastrointestinal disorders) | 3 | 7 | 12
Abdominal pain (Gastrointestinal disorders) | 1 | 5 | 6
Oral disorder (Gastrointestinal disorders) | 3 | 3 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 4 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 5 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 1
Oral pain (Gastrointestinal disorders) | 1 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 2
Tongue ulceration (Gastrointestinal disorders) | 1 | 2 | 0
Toothache (Gastrointestinal disorders) | 1 | 2 | 0
Faeces discoloured (Gastrointestinal disorders) | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 8 | 15 | 14
Oedema peripheral (General disorders) | 6 | 7 | 7
Pyrexia (General disorders) | 3 | 9 | 8
Asthenia (General disorders) | 4 | 7 | 3
Chills (General disorders) | 3 | 5 | 2
Injection site erythema (General disorders) | 0 | 4 | 6
Injection site reaction (General disorders) | 0 | 3 | 6
Injection site pain (General disorders) | 0 | 7 | 1
Pain (General disorders) | 0 | 4 | 3
Mucosal inflammation (General disorders) | 1 | 4 | 1
Device occlusion (General disorders) | 1 | 1 | 2
Injection site bruising (General disorders) | 0 | 1 | 3
Injection site irritation (General disorders) | 0 | 2 | 2
Non-cardiac chest pain (General disorders) | 1 | 1 | 2
Catheter site pain (General disorders) | 0 | 0 | 2
Face oedema (General disorders) | 0 | 2 | 0
Facial pain (General disorders) | 0 | 2 | 0
Gait disturbance (General disorders) | 0 | 2 | 0
Generalised oedema (General disorders) | 1 | 1 | 0
Injection site discomfort (General disorders) | 0 | 0 | 2
Localised oedema (General disorders) | 1 | 1 | 0
Malaise (General disorders) | 0 | 0 | 2
Mucosal haemorrhage (General disorders) | 1 | 1 | 0
Oedema (General disorders) | 0 | 0 | 2
Feeling abnormal (General disorders) | 1 | 0 | 0
Local swelling (General disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 12 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 16 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Weight decreased (Investigations) | 5 | 15 | 10
Neutrophil count decreased (Investigations) | 0 | 5 | 4
White blood cell count decreased (Investigations) | 0 | 4 | 5
Platelet count decreased (Investigations) | 0 | 6 | 2
Alanine aminotransferase increased (Investigations) | 1 | 5 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 5 | 1
Blood magnesium decreased (Investigations) | 1 | 4 | 0
Blood creatinine increased (Investigations) | 1 | 2 | 1
Cardiac murmur (Investigations) | 3 | 1 | 0
International normalised ratio increased (Investigations) | 1 | 3 | 0
Lymphocyte count decreased (Investigations) | 1 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 2 | 1
Transaminases increased (Investigations) | 2 | 1 | 0
Weight increased (Investigations) | 1 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 2 | 0
Staphylococcus test positive (Investigations) | 1 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 2
Activated partial thromboplastin time abnormal (Investigations) | 1 | 0 | 0
Clostridium test positive (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 4 | 4
Cellulitis (Infections and infestations) | 1 | 5 | 4
Urinary tract infection (Infections and infestations) | 1 | 3 | 6
Upper respiratory tract infection (Infections and infestations) | 0 | 6 | 3
Herpes simplex (Infections and infestations) | 2 | 4 | 1
Oral candidiasis (Infections and infestations) | 2 | 2 | 3
Herpes zoster (Infections and infestations) | 1 | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 2 | 2
Respiratory tract infection (Infections and infestations) | 0 | 4 | 0
Sinusitis (Infections and infestations) | 0 | 3 | 1
Fungal infection (Infections and infestations) | 1 | 1 | 1
Furuncle (Infections and infestations) | 0 | 3 | 0
Hordeolum (Infections and infestations) | 0 | 2 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 2
Rash pustular (Infections and infestations) | 1 | 2 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 2
Ear infection (Infections and infestations) | 1 | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 2 | 0
Osteomyelitis (Infections and infestations) | 0 | 2 | 0
Tooth infection (Infections and infestations) | 0 | 2 | 0
Body tinea (Infections and infestations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 18 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 12 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 8 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 5 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 2 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 5 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin K deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 11 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 11 | 11
Neutropenia (Blood and lymphatic system disorders) | 4 | 6 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 6 | 2
Pancytopenia (Blood and lymphatic system disorders) | 2 | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Spleen disorder (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenic lesion (Blood and lymphatic system disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 14 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 10 | 6
Erythema (Skin and subcutaneous tissue disorders) | 0 | 7 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 3 | 4 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 2 | 4 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 4 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 8 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 7 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 7 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 12 | 6
Headache (Nervous system disorders) | 1 | 9 | 4
Dysgeusia (Nervous system disorders) | 1 | 6 | 3
Syncope (Nervous system disorders) | 2 | 2 | 3
Tremor (Nervous system disorders) | 0 | 4 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 1
Balance disorder (Nervous system disorders) | 0 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 2 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 4 | 8 | 2
Anxiety (Psychiatric disorders) | 0 | 10 | 3
Depression (Psychiatric disorders) | 1 | 4 | 4
Confusional state (Psychiatric disorders) | 1 | 4 | 2
Agitation (Psychiatric disorders) | 1 | 2 | 2
Mental status changes (Psychiatric disorders) | 1 | 2 | 2
Delirium (Psychiatric disorders) | 0 | 3 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 5 | 1
Tachycardia (Cardiac disorders) | 1 | 2 | 5
Angina pectoris (Cardiac disorders) | 1 | 2 | 1
Bradycardia (Cardiac disorders) | 0 | 4 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 2
Atrial flutter (Cardiac disorders) | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 4 | 6 | 1
Hypertension (Vascular disorders) | 1 | 3 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 2 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 5 | 6
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 2
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 2
Wound (Injury, poisoning and procedural complications) | 0 | 2 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 3 | 4
Haematuria (Renal and urinary disorders) | 0 | 5 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 2 | 2
Urinary retention (Renal and urinary disorders) | 1 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 0
Renal cyst (Renal and urinary disorders) | 0 | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 2 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 2
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 2 | 2 | 1
Erythema of eyelid (Eye disorders) | 1 | 0 | 0
Eye inflammation (Eye disorders) | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Accrual to the lenalidomide arm was stopped before ending accrual to the 2 other arms because of poor tolerability and no comparison of outcomes was planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications